CLINICAL TRIAL: NCT02853331
Title: A Phase III Randomized, Open-label Study to Evaluate Efficacy and Safety of Pembrolizumab (MK-3475) in Combination With Axitinib Versus Sunitinib Monotherapy as a First-line Treatment for Locally Advanced or Metastatic Renal Cell Carcinoma (mRCC) (KEYNOTE-426)
Brief Title: Study to Evaluate the Efficacy and Safety of Pembrolizumab (MK-3475) in Combination With Axitinib Versus Sunitinib Monotherapy in Participants With Renal Cell Carcinoma (MK-3475-426/KEYNOTE-426)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-426; 163460 (Registry Identifier: JAPIC-CTI); MK-3475-426 (Other: MSD); KEYNOTE-426 (Other: MSD); 2023-507294-18-00 (Registry Identifier: EU CT); U1111-1295-6836 (Registry Identifier: UTN); 2016-000588-17 (EudraCT Number)
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Results first posted 2019-11-08 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: Renal Cell Carcinoma
Keywords: PD1; PD-1; PDL1; PD-L1; PDL2; PD-L2; VEGFR TKI
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pembrolizumab; Axitinib; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab+Axitinib Combination Therapy (Experimental): Participants receive pembrolizumab 200 mg intravenously every 3 weeks PLUS axitinib 5 mg orally twice daily.
  Interventions: Biological: Pembrolizumab; Drug: Axitinib
- Sunitinib Monotherapy (Active Comparator): Participants receive sunitinib 50 mg orally once daily for 4 weeks and then are off treatment for 2 weeks.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Biological: Pembrolizumab — Intravenous infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab+Axitinib Combination Therapy
Drug: Axitinib — Oral tablet
  Other Names: INLYTA®
  Arms: Pembrolizumab+Axitinib Combination Therapy
Drug: Sunitinib — Oral capsule
  Other Names: SUTENT®
  Arms: Sunitinib Monotherapy

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of pembrolizumab (MK-3475) in combination with axitinib versus sunitinib monotherapy as a first-line treatment for participants with advanced/metastatic renal cell carcinoma (mRCC).

The primary hypotheses of this study are:

1. The combination therapy of pembrolizumab plus axitinib is superior to sunitinib monotherapy with respect to Progression-Free Survival (PFS) as assessed by blinded independent central imaging review per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)
2. The combination therapy of pembrolizumab plus axitinib is superior to sunitinib monotherapy with respect to Overall Survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Has histologically confirmed diagnosis of RCC with clear cell component with or without sarcomatoid features
* Has locally advanced/metastatic disease (i.e., newly diagnosed Stage IV RCC per American Joint Committee on Cancer) or has recurrent disease
* Has measurable disease per RECIST 1.1 as assessed by the investigator/site radiologist
* Has received no prior systemic therapy for advanced RCC.
* Has provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated.
* Has Karnofsky performance status (KPS) ≥ 70% as assessed within 10 days prior to randomization.
* If receiving bone resorptive therapy (including but not limited to bisphosphonate or RANK-L inhibitor) must have therapy initiated at least 2 weeks prior to randomization.
* Demonstrates adequate organ function.
* Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study drug.
* Male participants of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study drug through 120 days after the last dose of study drug.

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to randomization.
* Has had major surgery within 4 weeks, received radiation therapy within 2 weeks prior to randomization, or has not recovered (i.e., ≤ Grade 1 or at baseline) from AEs due to prior treatment.
* Has had prior treatment with any anti-programmed cell death (anti-PD-1), or programmed cell death ligand 1 (PD-L1), or PD-L2 agent or an antibody targeting any other immune-regulatory receptors or mechanisms.
* Has received prior systemic anti-cancer therapy for RCC with vascular endothelial growth factor (VEGF)/VEGF receptors (VEGFR) or mechanistic target of rapamycin (mTOR) targeting agents.
* Has a history of severe hypersensitivity reaction (e.g., generalized rash/erythema, hypotension, bronchospasm, angioedema or anaphylaxis) to axitinib or sunitinib.
* Has a diagnosis of immunodeficiency OR is receiving a systemic steroid therapy exceeding physiologic corticosteroid dose or any other form of immunosuppressive therapy within 7 days prior to randomization, except in the case of central nervous system (CNS) metastases.
* Has an active autoimmune disease requiring systemic treatment with in the past 2 years OR a documented history of clinically severe autoimmune disease. Note: Participants with vitiligo, Sjøgren's syndrome, Type 1 diabetes, resolved childhood asthma/atopy, hypothyroidism or adrenal or pituitary insufficiency who are stable on hormone replacement, are not excluded.
* Has a known additional malignancy that has progressed or has required active treatment in the last 3 years. Note: Basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ such as breast cancer in situ are acceptable if they have undergone potentially curative therapy.
* Has known active CNS metastases and/or carcinomatous meningitis.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV).
* Has known active Hepatitis B or Hepatitis C infection.
* Has received a live virus vaccine within 30 days of randomization.
* Has a clinically significant gastrointestinal (GI) abnormality including:
* Malabsorption, total gastric resection
* Or any condition that might affect the absorption of orally taken medication
* Active GI bleeding, as evidenced by hematemesis, hematochezia or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy
* Intraluminal metastatic lesion with suspected bleeding, inflammatory bowel disease, ulcerative colitis or other GI condition associated with increased risk of perforation
* Has QT interval corrected for heart rate (QTc) ≥480 msec.
* Has a history of any of the following cardiovascular conditions within 12 months of randomization:
* Myocardial infarction
* Unstable angina pectoris
* Cardiac angioplasty or stenting
* Coronary/peripheral artery bypass graft
* Class III or IV congestive heart failure per New York Heart Association
* Cerebrovascular accident or transient ischemic attack
* Has a history of deep vein thrombosis or pulmonary embolism within 6 months of screening.
* Has poorly controlled hypertension defined as systolic blood pressure (SBP) ≥150 mm Hg and/or diastolic blood pressure (DBP) ≥90 mm Hg.
* Has evidence of inadequate wound healing.
* Has active bleeding disorder or other history of significant bleeding episodes within 30 days of randomization.
* Has hemoptysis within 6 weeks prior to randomization.
* Has current use (within 7 days of randomization) or anticipated need for treatment with drugs or foods that are known strong cytochrome P450 (CYP3A4/5) inhibitors.
* Has current use (within 7 days of randomization) or anticipated need for treatment with drugs that are known strong CYP3A4/5 inducers, including but not limited to carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, and St. John's wort; or drugs that are known with proarrhythmic potential.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Has had a prior solid organ transplant.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 861 (Actual)
Dates: Start 2016-09-16 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2025-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Rini BI, Plimack ER, Stus V, Gafanov R, Waddell T, Nosov D, Pouliot F, Alekseev B, Soulieres D, Melichar B, Vynnychenko I, de Azevedo SJ, Borchiellini D, McDermott RS, Bedke J, Tamada S, Wu S, Markensohn J, Zhang Y, Loboda A, Vajdi A, Perini RF, Burgents J, Powles T. Pembrolizumab plus axitinib versus sunitinib for advanced clear cell renal cell carcinoma: 5-year survival and biomarker analyses of the phase 3 KEYNOTE-426 trial. Nat Med. 2025 Oct;31(10):3475-3484. doi: 10.1038/s41591-025-03867-5. Epub 2025 Aug 1. PMID 40750932
- [Derived] Chung HJ, Kondoh C, Bae WK, Tamada S, Matsubara N, Lee HJ, Mizuno R, Anai S, Kimura G, Tomita Y, Chang CH, Chang JW, Lin J, Perini RF, Molife LR, Powles T, Rini BI, Uemura H. First-line pembrolizumab-axitinib versus sunitinib in metastatic RCC: subgroup analysis of patients enrolled in the phase 3 KEYNOTE-426 in Eastern Asia. Jpn J Clin Oncol. 2025 Apr 6;55(4):406-413. doi: 10.1093/jjco/hyae182. PMID 39815637
- [Derived] Rini BI, Atkins MB, Choueiri TK, Teresi RE, Rosbrook B, Thakur M, Hutson TE. Plain language summary looking at how long side effects last after treatment with axitinib is stopped in people with advanced renal cell carcinoma. Future Oncol. 2023 Dec;19(40):2623-2629. doi: 10.2217/fon-2023-0233. Epub 2023 Aug 1. PMID 37526095
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Bedke J, Rini BI, Plimack ER, Stus V, Gafanov R, Waddell T, Nosov D, Pouliot F, Soulieres D, Melichar B, Vynnychenko I, Azevedo SJ, Borchiellini D, McDermott RS, Tamada S, Nguyen AM, Wan S, Perini RF, Rhoda Molife L, Atkins MB, Powles T. Health-related Quality of Life Analysis from KEYNOTE-426: Pembrolizumab plus Axitinib Versus Sunitinib for Advanced Renal Cell Carcinoma. Eur Urol. 2022 Oct;82(4):427-439. doi: 10.1016/j.eururo.2022.06.009. Epub 2022 Jul 15. PMID 35843776
- [Derived] Rini BI, Atkins MB, Plimack ER, Soulieres D, McDermott RS, Bedke J, Tartas S, Alekseev B, Melichar B, Shparyk Y, Kondoh C, Langiewicz P, Wood LA, Hammers H, Silber CG, Haber B, Jensen E, Chen M, Powles T. Characterization and Management of Treatment-emergent Hepatic Toxicity in Patients with Advanced Renal Cell Carcinoma Receiving First-line Pembrolizumab plus Axitinib. Results from the KEYNOTE-426 Trial. Eur Urol Oncol. 2022 Apr;5(2):225-234. doi: 10.1016/j.euo.2021.05.007. Epub 2021 Jul 6. PMID 34244116
- [Derived] Rini BI, Atkins MB, Choueiri TK, Thomaidou D, Rosbrook B, Thakur M, Hutson TE. Time to Resolution of Axitinib-Related Adverse Events After Treatment Interruption in Patients With Advanced Renal Cell Carcinoma. Clin Genitourin Cancer. 2021 Oct;19(5):e306-e312. doi: 10.1016/j.clgc.2021.03.019. Epub 2021 Apr 5. PMID 33947608
- [Derived] Powles T, Plimack ER, Soulieres D, Waddell T, Stus V, Gafanov R, Nosov D, Pouliot F, Melichar B, Vynnychenko I, Azevedo SJ, Borchiellini D, McDermott RS, Bedke J, Tamada S, Yin L, Chen M, Molife LR, Atkins MB, Rini BI. Pembrolizumab plus axitinib versus sunitinib monotherapy as first-line treatment of advanced renal cell carcinoma (KEYNOTE-426): extended follow-up from a randomised, open-label, phase 3 trial. Lancet Oncol. 2020 Dec;21(12):1563-1573. doi: 10.1016/S1470-2045(20)30436-8. Epub 2020 Oct 23. PMID 33284113
- [Derived] Rini BI, Plimack ER, Stus V, Gafanov R, Hawkins R, Nosov D, Pouliot F, Alekseev B, Soulieres D, Melichar B, Vynnychenko I, Kryzhanivska A, Bondarenko I, Azevedo SJ, Borchiellini D, Szczylik C, Markus M, McDermott RS, Bedke J, Tartas S, Chang YH, Tamada S, Shou Q, Perini RF, Chen M, Atkins MB, Powles T; KEYNOTE-426 Investigators. Pembrolizumab plus Axitinib versus Sunitinib for Advanced Renal-Cell Carcinoma. N Engl J Med. 2019 Mar 21;380(12):1116-1127. doi: 10.1056/NEJMoa1816714. Epub 2019 Feb 16. PMID 30779529
- [Derived] Atkins MB, Plimack ER, Puzanov I, Fishman MN, McDermott DF, Cho DC, Vaishampayan U, George S, Olencki TE, Tarazi JC, Rosbrook B, Fernandez KC, Lechuga M, Choueiri TK. Axitinib in combination with pembrolizumab in patients with advanced renal cell cancer: a non-randomised, open-label, dose-finding, and dose-expansion phase 1b trial. Lancet Oncol. 2018 Mar;19(3):405-415. doi: 10.1016/S1470-2045(18)30081-0. Epub 2018 Feb 10. PMID 29439857
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26260&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: These interim results are based on a database cutoff date of 24-Aug-2018, at which time 693 participants were ongoing in the study.
Groups:
- Pembrolizumab + Axitinib: Participants received pembrolizumab 200 mg intravenously every 3 weeks PLUS axitinib 5 mg orally twice daily.
- Sunitinib: Participants received sunitinib 50 mg orally once daily for 4 weeks and then were off treatment for 2 weeks.
Period: Overall Study
Arm/Group | Pembrolizumab + Axitinib | Sunitinib
Started | 432 | 429
Treated | 429 | 425
Completed | 0 | 0
Not Completed | 432 | 429
Not completed — Death | 59 | 95
Not completed — Withdrawal by Subject | 5 | 9
Not completed — Ongoing in study | 368 | 325

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Axitinib | Sunitinib | Total
Number analyzed (Participants) | 432 | 429 | 861
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.2 (10.0) | 60.8 (10.2) | 61.0 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 109 | 233
  Male | 308 | 320 | 628
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 18 | 37
  Not Hispanic or Latino | 377 | 387 | 764
  Unknown or Not Reported | 36 | 24 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 66 | 71 | 137
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 8 | 18
  White | 343 | 341 | 684
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 9 | 22
International Metastatic Renal Cell Carcinoma Database Consortium (IMDC) Risk Group [Count of Participants; unit: Participants] — Participants were stratified by IMDC risk group using the following criteria: baseline Karnofsky Performance Status <80%; interval between initial diagnosis of renal cell carcinoma to start of first-line systemic treatment for advanced disease <1year; baseline hemoglobin <lower limit of normal (LLN); baseline platelet count >upper limit of normal (ULN); baseline corrected calcium1 >ULN; and baseline neutrophil >ULN. The category was determined by totaling the risk factors per participant and scored as favorable (no factors); intermediate (1 or 2 factors); and poor (≥3 factors).
  Participants
    Favorable | 138 | 131 | 269
    Intermediate | 238 | 246 | 484
    Poor | 56 | 52 | 108
Geographic Region [Count of Participants; unit: Participants] — Participants were stratified by geographic region using the following categories: North America; Western Europe; and Rest of the World.
  Participants
    North America | 104 | 103 | 207
    Western Europe | 106 | 104 | 210
    Rest of World | 222 | 222 | 444

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Imaging Review
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The PFS per RECIST 1.1 was calculated using the product-limit (Kaplan-Meier) method for censored data. The PFS for participants is presented.
Time Frame: Through Database Cutoff Date of 24-Aug-2018 (up to approximately 22 months)
Population: The analysis population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Axitinib | Sunitinib
Number analyzed (Participants) | 432 | 429
Months | 15.1 [12.6 to 17.7] | 11.0 [8.7 to 12.5]
Statistical Analysis 1: Comparison: Pembrolizumab + Axitinib vs Sunitinib; Test type: Superiority; p = 0.00012, Log Rank; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.56 to 0.84] — HR based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by IMDC risk group (favorable vs. intermediate vs. poor) and geographic region (North America vs. Western Europe vs. Rest of World)

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the interim analysis were censored at the date of the last follow up. The OS was calculated using the product-limit (Kaplan-Meier) method for censored data. The OS for participants is presented.
Time Frame: Through Database Cutoff Date of 24-Aug-2018 (up to approximately 22 months)
Population: The analysis population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Axitinib | Sunitinib
Number analyzed (Participants) | 432 | 429
Months | NA [NA to NA] — OS median, OS lower limit & OS upper limit were not reached by the time of the data cutoff (24-Aug-2018). | NA [NA to NA] — OS median, OS lower limit & OS upper limit were not reached by the time of the data cutoff (24-Aug-2018).
Statistical Analysis 1: Comparison: Pembrolizumab + Axitinib vs Sunitinib; Test type: Superiority; p = 0.00005, Log Rank; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.38 to 0.74] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Imaging Review
Description: ORR was determined per RECIST 1.1 and was defined as the percentage of participants in the analysis population who had a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1. The ORR was calculated using the Miettinen & Nurminen method stratified by International Metastatic Renal Cell Carcinoma (RCC) Database Consortium (IMDC) risk group (favorable vs. intermediate vs. poor) and geographic region (North America vs. Western Europe vs. Rest of World). The percentage of participants who experienced a CR or PR is presented.
Time Frame: Through Database Cutoff Date of 24-Aug-2018 (up to approximately 22 months)
Population: The analysis population consisted of all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Axitinib | Sunitinib
Number analyzed (Participants) | 432 | 429
Percentage of participants | 59.3 [54.5 to 63.9] | 35.7 [31.1 to 40.4]
Statistical Analysis 1: Comparison: Pembrolizumab + Axitinib vs Sunitinib; Test type: Superiority; p < 0.0001, Miettinen & Nurminen method; H0: difference in %=0 versus H1: difference in % >0; Difference in percentages = 23.6, 95% CI 2-sided [17.2 to 29.9] — Difference in percentages based on Miettinen & Nurminen method stratified by IMDC risk group (favorable vs. intermediate vs. poor) and geographic region (North America vs. Western Europe vs. Rest of World)

4. Secondary Outcome: Disease Control Rate (DCR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Imaging Review
Description: DCR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions), Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters), or Stable Disease (SD) per RECIST 1.1 for ≥6 months. The DCR was calculated using the Miettinen & Nurminen method stratified by International Metastatic Renal Cell Carcinoma (RCC) Database Consortium (IMDC) risk group (favorable vs. intermediate vs. poor) and geographic region (North America vs. Western Europe vs. Rest of World). The percentage of participants who experienced a CR, PR, or SD is presented.
Time Frame: Through Database Cutoff Date of 24-Aug-2018 (up to approximately 22 months)
Population: The analysis population consisted of all randomized participants who experienced a PR, CR or SD for ≥6 months.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Axitinib | Sunitinib
Number analyzed (Participants) | 432 | 429
Percentage of participants | 71.5 [67.0 to 75.7] | 60.6 [55.8 to 65.3]
Statistical Analysis 1: Comparison: Pembrolizumab + Axitinib vs Sunitinib; Test type: Superiority; Difference in percentages = 11.0, 95% CI 2-sided [4.8 to 17.0] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Duration of Response (DOR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Imaging Review
Description: DOR was defined as the time from first documented evidence of a Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1 until progressive disease (PD) or death due to any cause, whichever occurred first. PD was defined per RECIST 1.1 as ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The DOR was calculated using the product-limit (Kaplan-Meier) method for censored data. The DOR for all participants who experienced a CR or PR is presented.
Time Frame: Through Database Cutoff Date of 24-Aug-2018 (up to approximately 22 months)
Population: The analysis population consisted of all randomized participants who experienced a CR or PR.
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab + Axitinib | Sunitinib
Number analyzed (Participants) | 256 | 153
Months | NA [1.4 to NA] — Median DOR not reached by the time of the data cutoff (24-Aug-2018). DOR upper limit not calculated due to no progressive disease by the time of last disease assessment. | 15.2 [1.1 to NA] — DOR upper limit not calculated due to no progressive disease by the time of last disease assessment.

6. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of study treatment, was also an AE. The number of participants who experienced at least one AE is presented.
Time Frame: Through Database Cutoff Date of 24-Aug-2018 (up to approximately 22 months)
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Axitinib | Sunitinib
Number analyzed (Participants) | 429 | 425
Participants | 422 | 423

7. Secondary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of study treatment, was also an AE. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Through Database Cutoff Date of 24-Aug-2018 (up to approximately 22 months)
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Axitinib | Sunitinib
Number analyzed (Participants) | 429 | 425
Participants | 131 | 59

8. Secondary Outcome: Progression Free Survival Rate (PFS Rate) at Month 12 in All Participants
Description: The PFS rate was determined in all participants at Month 12. PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1), PD was defined as ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The date of PD was approximated by the date of the first assessment at which PD was documented per RECIST 1.1 by Blinded Independent Central Review (BICR). Death was always considered as confirmed PD. Participants who did not experience PFS were censored at the last disease assessment. The PFS rate at Month 12 is presented.
Time Frame: Month 12
Population: The analysis population consisted of all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Axitinib | Sunitinib
Number analyzed (Participants) | 432 | 429
Percentage of participants | 59.6 [54.3 to 64.5] | 46.1 [40.5 to 51.5]

9. Secondary Outcome: Progression Free Survival Rate (PFS Rate) at Month 18 in All Participants
Description: The PFS rate was determined in all participants at Month 18. PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1), PD was defined as ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The date of PD was approximated by the date of the first assessment at which PD was documented per RECIST 1.1 by Blinded Independent Central Review (BICR). Death was always considered as confirmed PD. Participants who did not experience PFS were censored at the last disease assessment. The PFS rate at Month 18 is presented.
Time Frame: Month 18
Population: The analysis population consisted of all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Axitinib | Sunitinib
Number analyzed (Participants) | 432 | 429
Percentage of participants | 41.1 [33.5 to 48.5] | 32.8 [25.4 to 40.4]

10. Secondary Outcome: Progression Free Survival Rate (PFS Rate) at Month 24 in All Participants
Description: The PFS rate was determined in all participants at Month 24. PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1), PD was defined as ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The date of PD was approximated by the date of the first assessment at which PD was documented per RECIST 1.1 by Blinded Independent Central Review (BICR). Death was always considered as confirmed PD. Participants who did not experience PFS were censored at the last disease assessment.
Time Frame: Month 24
Reporting Status: Not Posted, anticipated posting 2026-12

11. Secondary Outcome: Overall Survival (OS) Rate at Month 12 in All Participants
Description: The OS rate was determined for all participants at Month 12 and was defined as the time from randomization to death due to any cause. Participants were censored at the date of their last assessment. The OS rate at Month 12 is presented.
Time Frame: Month 12
Population: The analysis population consisted of all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Axitinib | Sunitinib
Number analyzed (Participants) | 432 | 429
Percentage of participants | 89.9 [86.4 to 92.4] | 78.3 [73.8 to 82.1]

12. Secondary Outcome: Overall Survival (OS) Rate at Month 18 in All Participants
Description: The OS rate was determined for all participants at Month 18 and was defined as the time from randomization to death due to any cause. Participants were censored at the date of their last assessment. The OS rate at Month 18 is presented.
Time Frame: Month 18
Population: The analysis population consisted of all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Axitinib | Sunitinib
Number analyzed (Participants) | 432 | 429
Percentage of participants | 82.3 [77.2 to 86.3] | 72.1 [66.3 to 77.0]

13. Secondary Outcome: Overall Survival (OS) Rate at Month 24 in All Participants
Description: The OS rate was determined for all participants at Month 24 and was defined as the time from randomization to death due to any cause. Participants were censored at the date of their last assessment.
Time Frame: Month 24
Reporting Status: Not Posted, anticipated posting 2026-12

14. Secondary Outcome: Time to True Deterioration (TTD) of the Functional Assessment of Cancer Therapy Kidney Symptom Index Disease-Related Symptoms (FKSI-DRS) Score
Description: TTD was defined as time (in months) from the first dose of study treatment to the date of deterioration of FKSI-DRS Score. The FKSI-DRS was a questionnaire that asked the participant to rate 9 kidney cancer-related symptoms: lack of energy, fatigue, weight loss, pain, bone pain, shortness of breath, cough, fever, or blood in the urine. Each item was scored on a 5-point scale (0=not at all to 4=very much). FKSI-DRS total score ranged from 0 (most severe symptoms) to 36 (no symptoms) with a higher score indicating a better outcome. Deterioration was defined as a 3-point decrease (i.e. lower score) in symptom score and the time to true deterioration was the time to first onset of 3 or more decreases from baseline with confirmation under right-censoring rule (the last observation). The time to true deterioration as measured in months is presented.
Time Frame: Through Database Cutoff Date of 24-Aug-2018 (up to approximately 22 months)
Population: All randomized participants who received at least 1 dose of study medication and completed at least 1 questionnaire assessment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Axitinib | Sunitinib
Number analyzed (Participants) | 395 | 387
Months | NA [12.7 to NA] — TTD median not reached by the time of the data cutoff (24-Aug-2018). For TTD upper limit, no deterioration reached by the time of last disease assessment. | NA [NA to NA] — TTD median not reached by the time of the data cutoff (24-Aug-2018). For TTD lower and upper limit, no deterioration reached by the time of last disease assessment.

15. Secondary Outcome: Least Squares (LS) Mean Change From Baseline to Week 54 in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status (GHS) Scale Score
Description: EORTC QLQ-C30 is a questionnaire that rates the overall quality of life in cancer participants. The first 28 questions use a 4-point scale (1=not at all to 4=very much) for evaluating function (physical, role, social, cognitive, emotional), symptoms (diarrhea, fatigue, dyspnea, appetite loss, insomnia, nausea/vomiting, constipation, and pain) and financial difficulties. The last 2 questions use a 7-point scale (1=very poor to 7=excellent) to evaluate overall health and quality of life. Global scores are converted to a score of 0 to 100, with a higher score indicating improved health status.
Time Frame: Baseline (prior to first dose of study treatment in Cycle 1 [cycle length = 21 days]) and Week 54
Reporting Status: Not Posted, anticipated posting 2026-12

16. Other Pre Specified Outcome: Mean Baseline EORTC Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Score
Description: EORTC QLQ-C30 is a questionnaire that rates the overall quality of life in cancer participants. The first 28 questions use a 4-point scale (1=not at all to 4=very much) for evaluating function (physical, role, social, cognitive, emotional), symptoms (diarrhea, fatigue, dyspnea, appetite loss, insomnia, nausea/vomiting, constipation, and pain) and financial difficulties. The last 2 questions use a 7-point scale (1=very poor to 7=excellent) to evaluate overall health and quality of life. Global scores are converted to a score of 0 to 100, with a higher score indicating improved health status. The mean baseline EORTC QLQ-C30 score is presented.
Time Frame: Baseline (prior to first dose of study treatment in Cycle 1 [cycle length = 21 days])
Population: All participants with non-missing questionnaire assessments at baseline.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pembrolizumab + Axitinib | Sunitinib
Number analyzed (Participants) | 394 | 410
Score on a scale | 70.90 (21.037) | 72.07 (20.642)

17. Post Hoc Outcome: Least Squares (LS) Mean Change From Baseline to Week 30 in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status (GHS) Scale Score
Description: EORTC QLQ-C30 is a cancer-specific instrument with 30 questions used to assess the overall quality of life (QOL) in cancer participants. The first 28 questions used a 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much) for evaluating 5 functional scales (physical, role, social, cognitive, emotional), 8 symptom scales/items (diarrhea, fatigue, dyspnea, appetite loss, insomnia, nausea and vomiting [N/V], constipation, and pain) and a single item (financial difficulties). The last 2 questions represented the participant's assessment of overall health and quality of life on a 7-point scale (1=very poor to 7=excellent). EORTC QLQ-C30 global scores were linearly transformed on a scale of 0 to 100; with a high score indicating improved health status. Negative change from baseline values indicated deterioration in health status or functioning and positive changes indicated improvement. The LS Mean change from baseline to Week 30 is presented.
Time Frame: Baseline (prior to first dose of study treatment in Cycle 1 [cycle length = 21 days]) and Week 30
Population: All participants who received at least 1 dose of study medication and had non-missing questionnaire assessments at baseline and Week 30.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Axitinib | Sunitinib
Number analyzed (Participants) | 427 | 423
Score on a scale | -4.05 [-6.03 to -2.07] | -2.35 [-4.44 to -0.26]

ADVERSE EVENTS:
Time Frame: Through Database Cutoff Date of 24-Aug-2018 (up to approximately 22 months)
Description: Population: All participants who received ≥1 dose of study treatment. Per protocol, progression of cancer under study was not considered an AE unless related to study drug. Therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study drug are excluded as AEs.
Arm/Group | Pembrolizumab + Axitinib | Sunitinib
All-Cause Mortality (participants affected / at risk) | 59/432 | 97/429
Serious Adverse Events (participants affected / at risk) | 173/429 | 133/425
Other Adverse Events (participants affected / at risk) | 417/429 | 415/425
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Axitinib (N=429) | Sunitinib (N=425)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac amyloidosis (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (3)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 4 (4) | 0 (0)
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Hypophysitis (Endocrine disorders) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 2 (2)
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 12 (12) | 4 (4)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Asthenia (General disorders) | 3 (3) | 4 (4)
Chest pain (General disorders) | 2 (2) | 1 (1)
Condition aggravated (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 3 (3)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 2 (2)
Malaise (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (3)
Pyrexia (General disorders) | 3 (3) | 1 (1)
Strangulated hernia (General disorders) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 5 (5) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Hepatitis fulminant (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 3 (3) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0)
Contrast media reaction (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Acute hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Extrapulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 1 (1)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pancreas infection (Infections and infestations) | 1 (1) | 0 (0)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (2)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 10 (12)
Sepsis (Infections and infestations) | 1 (1) | 2 (3)
Skin infection (Infections and infestations) | 0 (0) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (4) | 3 (3)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 6 (6) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood electrolytes abnormal (Investigations) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 2 (2) | 0 (0)
Liver function test increased (Investigations) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 3 (3)
Transaminases increased (Investigations) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 6 (7) | 5 (5)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 4 (4) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (2)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (4) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 4 (4) | 0 (0)
Pachymeningitis (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Dependence (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 7 (8) | 3 (3)
Calculus urinary (Renal and urinary disorders) | 2 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (7)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 2 (2)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Axitinib (N=429) | Sunitinib (N=425)
Anaemia (Blood and lymphatic system disorders) | 32 (34) | 97 (152)
Leukopenia (Blood and lymphatic system disorders) | 6 (11) | 41 (79)
Neutropenia (Blood and lymphatic system disorders) | 8 (11) | 82 (152)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (13) | 95 (164)
Hyperthyroidism (Endocrine disorders) | 53 (58) | 16 (18)
Hypothyroidism (Endocrine disorders) | 152 (177) | 133 (172)
Abdominal pain (Gastrointestinal disorders) | 48 (64) | 29 (32)
Abdominal pain upper (Gastrointestinal disorders) | 26 (35) | 26 (31)
Constipation (Gastrointestinal disorders) | 89 (107) | 62 (70)
Diarrhoea (Gastrointestinal disorders) | 231 (496) | 191 (380)
Dry mouth (Gastrointestinal disorders) | 25 (27) | 25 (26)
Dyspepsia (Gastrointestinal disorders) | 22 (26) | 62 (73)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 18 (18) | 48 (60)
Nausea (Gastrointestinal disorders) | 119 (174) | 134 (205)
Stomatitis (Gastrointestinal disorders) | 67 (86) | 88 (110)
Vomiting (Gastrointestinal disorders) | 64 (97) | 78 (125)
Asthenia (General disorders) | 62 (85) | 60 (77)
Fatigue (General disorders) | 165 (208) | 158 (211)
Mucosal inflammation (General disorders) | 56 (77) | 92 (143)
Oedema peripheral (General disorders) | 28 (29) | 34 (43)
Pyrexia (General disorders) | 53 (65) | 42 (46)
Nasopharyngitis (Infections and infestations) | 33 (41) | 15 (23)
Upper respiratory tract infection (Infections and infestations) | 27 (31) | 20 (20)
Urinary tract infection (Infections and infestations) | 37 (54) | 25 (28)
Alanine aminotransferase increased (Investigations) | 110 (158) | 64 (81)
Aspartate aminotransferase increased (Investigations) | 108 (163) | 69 (95)
Blood alkaline phosphatase increased (Investigations) | 27 (32) | 19 (21)
Blood bilirubin increased (Investigations) | 28 (45) | 24 (39)
Blood creatinine increased (Investigations) | 48 (79) | 51 (72)
Blood thyroid stimulating hormone increased (Investigations) | 23 (25) | 22 (28)
Neutrophil count decreased (Investigations) | 4 (6) | 50 (109)
Platelet count decreased (Investigations) | 16 (21) | 76 (148)
Weight decreased (Investigations) | 76 (86) | 47 (54)
White blood cell count decreased (Investigations) | 2 (2) | 43 (97)
Decreased appetite (Metabolism and nutrition disorders) | 126 (173) | 125 (156)
Hyperglycaemia (Metabolism and nutrition disorders) | 31 (53) | 20 (26)
Hyperkalaemia (Metabolism and nutrition disorders) | 30 (62) | 14 (16)
Hypophosphataemia (Metabolism and nutrition disorders) | 9 (20) | 36 (57)
Arthralgia (Musculoskeletal and connective tissue disorders) | 78 (95) | 25 (33)
Back pain (Musculoskeletal and connective tissue disorders) | 55 (64) | 42 (45)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 26 (29) | 18 (19)
Myalgia (Musculoskeletal and connective tissue disorders) | 36 (41) | 19 (23)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 51 (69) | 42 (48)
Dizziness (Nervous system disorders) | 22 (25) | 28 (31)
Dysgeusia (Nervous system disorders) | 47 (52) | 131 (185)
Headache (Nervous system disorders) | 67 (91) | 68 (87)
Insomnia (Psychiatric disorders) | 36 (40) | 39 (39)
Haematuria (Renal and urinary disorders) | 22 (23) | 20 (27)
Proteinuria (Renal and urinary disorders) | 74 (104) | 47 (77)
Cough (Respiratory, thoracic and mediastinal disorders) | 91 (108) | 58 (66)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 109 (126) | 14 (18)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 69 (80) | 44 (49)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 27 (30) | 40 (45)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 28 (31) | 19 (27)
Dry skin (Skin and subcutaneous tissue disorders) | 29 (31) | 39 (47)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 118 (140) | 169 (235)
Pruritus (Skin and subcutaneous tissue disorders) | 65 (78) | 25 (33)
Rash (Skin and subcutaneous tissue disorders) | 61 (84) | 47 (60)
Hypertension (Vascular disorders) | 189 (317) | 192 (278)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/31/NCT02853331/Prot_SAP_000.pdf